CLINICAL TRIAL: NCT01154010
Title: PEMF an Adjunct Therapy for Anterior Uveitis
Brief Title: PEMF: an Adjunct Therapy for Anterior Uveitis
Acronym: PEMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: BioElectronics Corporation (Industry)
Responsible Party: Principal Investigator, George Papaliodis, Director, Ocular Immunology and Uveitis Service, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 09-03-020
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: Anterior Uveitis; Iritis
Keywords: PEMF; iritis; anterior uveitis
MeSH Terms: conditions — Uveitis, Anterior; Iritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Device (Active Comparator): ActiPatch, a device that emits a low frequency energy called "pulsed electromagnetic field" (PEMF), will be worn by patients over the eye with anterior uveitis for 8 hours/day for 7 days. Patients will also be treated with topical steroids.
  Interventions: Device: PEMF
- Placebo Device (Placebo Comparator): Patients wear the PEMF placebo device for 8 hours/day for 7 days over the eye being treated for anterior uveitis. Patients will also be treated with topical steroids.
  Interventions: Device: PEMF Placebo

INTERVENTIONS:
Device: PEMF — ActiPatch will be worn by patients over the eye with anterior uveitis for 8 hours/day for 7 days. Patients will also be treated with topical steroids.
  Arms: Active Device
Device: PEMF Placebo — Patients wear the placebo device for 8 hours/day for 7 days over the eye being treated for anterior uveitis. Patients will also be treated with topical steroids.
  Arms: Placebo Device

SUMMARY:
The purpose of this study is to determine if a medical device (ActiPatch) that emits a low frequency pulsed electromagnetic field (PEMF) will benefit patients with anterior uveitis. Anterior uveitis (aka iritis) is an inflammatory disease involving the front segment of the eye. This is a common cause of a painful red eye, and ActiPatch has been shown to be effective in treating tissue inflammation. The conventional treatment of iritis typically involves frequent administration of topical steroids which have their own inherent risks (development of cataracts and/or glaucoma). The purpose of this study is to determine if ActiPatch therapy can be used to shorten the length of time and/or quantity of steroids administered.

DETAILED DESCRIPTION:
Iritis is an inflammatory disease focused in the anterior chamber of the eye. The inflammation inside the eye can lead to a number of conditions that ultimately effect vision. These can include glaucoma, posterior synechiae, cystoid macular edema, and cataract. The standard treatment for the disease is drug therapy centered around the administration of corticosteroids. These are administered in the form of eye drops, and if necessary periocular/intraocular injections, or/and by systemic oral/IV administration. Unfortunately, the treatment with corticosteroids can similarly induce severe side effects including glaucoma and cataract formation. ActiPatch is a medical device that emits a low frequency pulsed electromagnetic field. This device has been shown to reduce inflammation and pain in a number of conditions, eg blepharoplasty (eyelid surgery). ActiPatch is FDA approved for use after blepharoplasty to reduce swelling, inflammation and pain. The treatment is not invasive, does not require additional medication, and side effects from ActiPatch and other PEMF devices have not been reported. The potential benefit of treating uveitis with ActiPatch is the potential to reduce the time and/or amount of steroid administration. This would benefit patients by reducing the risk of unwanted side effects of the corticosteroid treatment.

The benefit to society would be an improved treatment for anterior uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Human subjects who have been clinically diagnosed with anterior uveitis (iritis) but are in otherwise in good health will be recruited for the study. The age requirement will be a minimum of 18 yrs. We will recruit 24 patient for this study. Subjects will only be included who have been clinically diagnosed with anterior uveitis (noninfectious). Eligibility will be determined by the treating Ophthalmologist (principal investigator) for inclusion in the study.

Exclusion Criteria:

* Vulnerable subjects, as defined by the Institutional Review Board (IRB), will not be recruited for participation (This includes individuals under 18, pregnant women, prisoners, fetuses, patients mentally or physically unable to provide written informed consent).
* Other groups excluded include: patients with pacemakers and patients with ferromagnetic metal implants since these devices may be effected by the pulsed electromagnetic field.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Papaliodis, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
A forthcoming article will include a chart that will document individual participant data.

REFERENCES:
- [Background] McLeod KJ, Lee RC, Ehrlich HP. Frequency dependence of electric field modulation of fibroblast protein synthesis. Science. 1987 Jun 12;236(4807):1465-9. doi: 10.1126/science.3589667.
- [Background] Nicolle FV, Bentall RM. Use of radio-frequency pulsed energy in the control of postoperative reaction in blepharoplasty. Aesthetic Plast Surg. 1982;6(3):169-71. doi: 10.1007/BF01570638. PMID 7180721
- [Background] Lee JH, McLeod KJ. Morphologic responses of osteoblast-like cells in monolayer culture to ELF electromagnetic fields. Bioelectromagnetics. 2000 Feb;21(2):129-36. doi: 10.1002/(sici)1521-186x(200002)21:23.0.co;2-q. PMID 10653624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Analysis in process as of December, 2016.
Pre-assignment Details: Analysis in process as of December, 2016.
Groups:
- Active Device: ActiPatch, a device that emits a low frequency energy called "pulsed electromagnetic field" (PEMF), will be worn by patients over the eye with anterior uveitis for 8 hours/day for 7 days. Patients will also be treated with topical steroids.
  PEMF: ActiPatch will be worn by patients over the eye with anterior uveitis for 8 hours/day for 7 days. Patients will also be treated with topical steroids.
  Analysis in process as of December, 2016.
- Placebo Device: Patients wear the PEMF placebo device for 8 hours/day for 7 days over the eye being treated for anterior uveitis. Patients will also be treated with topical steroids.
  PEMF Placebo: Patients wear the placebo device for 8 hours/day for 7 days over the eye being treated for anterior uveitis. Patients will also be treated with topical steroids.
  Analysis in process as of December, 2016.
Period: Overall Study
Arm/Group | Active Device | Placebo Device
Started | 9 | 9
Completed | 9 | 8
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Device | Placebo Device | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.33 (12.808) | 40.22 (14.228) | 41.275 (13.576)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Inflammation Grade at Day 7
Description: Degree and grade of ocular inflammation based on Standard Uveitis Nomenclature will be assessed at initial visit, Day 3, and Day 7 of use of the PEMF device to assess if the PEMF device decreases the duration and severity of ocular inflammation when used as an adjunctive therapy for anterior uveitis. The results posted here are from day 7. The Standard Uveitis Nomenclature scale ranges from 0 to 4, with 0 indicating a minimal level of ocular inflammation and 4 indicating the maximal level of corneal inflammation.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Device | Placebo Device
Number analyzed (Participants) | 9 | 8
units on a scale | 0.625 (0.876) | 1.444 (1.130)

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- Active Device: ActiPatch, a device that emits a low frequency energy called "pulsed electromagnetic field" (PEMF), will be worn by patients over the eye with anterior uveitis for 8 hours/day for 7 days. Patients will also be treated with topical steroids.
  PEMF: ActiPatch will be worn by patients over the eye with anterior uveitis for 8 hours/day for 7 days. Patients will also be treated with topical steroids.
  Analysis on-going as of December, 2016.
- Placebo Device: Patients wear the PEMF placebo device for 8 hours/day for 7 days over the eye being treated for anterior uveitis. Patients will also be treated with topical steroids.
  PEMF Placebo: Patients wear the placebo device for 8 hours/day for 7 days over the eye being treated for anterior uveitis. Patients will also be treated with topical steroids.
  Analysis on-going as of December, 2016.
Arm/Group | Active Device | Placebo Device
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No